CLINICAL TRIAL: NCT01848470
Title: Evaluation of Safety, Tolerability and Pharmacokinetic Characteristics of Multiple Ascending Doses of CG400549 in Healthy Volunteers
Brief Title: Multiple Ascending Doses Study of CG400549
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CG400549-1-02
Record Dates: First submitted 2013-02-13; First posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
MeSH Terms: interventions — CG 400549

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- E1. CG400549 640mg (Experimental): CG400549 640mg BID on Day 1-5 and QD on Day 6 in the fed-state
  Interventions: Drug: CG400549 640mg
- E2: CG400549 320mg (Experimental): CG400549 320mg QD on Day 1-5 in the fed-state.
  Interventions: Drug: CG400549 320 mg
- E3: CG400549 640mg (Experimental): CG400549 640mg QD on Day 1-5 in the fed-state.
  Interventions: Drug: CG400549 640 mg
- E4: CG400549 960mg (Experimental): CG400549 960mg QD on Day 1-5 in the fed-state.
  Interventions: Drug: CG400549 960 mg
- P1 Placebo (Placebo Comparator): Placebo 640mg BID on Day 1-5 and QD on Day 6 in the fed-state
  Interventions: Drug: Placebo 640mg
- P2: Placebo 320mg (Placebo Comparator): Placebo 320mg QD on Day 1-5 in the fed-state
  Interventions: Drug: Placebo 320mg
- P3 Placebo 640mg (Placebo Comparator): Placebo 640mg QD on Day 1-5 in the fed-state.
  Interventions: Drug: placebo 960 mg
- P4: Placebo 960mg (Placebo Comparator): Placebo 960mg QD on Day 1-5 in the fed-state.
  Interventions: Drug: Placebo 640mg

INTERVENTIONS:
Drug: CG400549 640mg — multiple oral doses of 640 mg CG400549 (n=6) BID for 5 days (Days 1-5) and a final dose on Day 6 in the fed state
  Arms: E1. CG400549 640mg
Drug: CG400549 320 mg — multiple oral doses of 320 mg CG400549 (n=6) QD for 5 days in the fed state
  Arms: E2: CG400549 320mg
Drug: CG400549 640 mg — multiple oral doses of 640 mg CG400549 (n=6) QD for 5 days in the fed state
  Arms: E3: CG400549 640mg
Drug: CG400549 960 mg — multiple oral doses of 960 mg CG400549 (n=6) QD for 5 days in the fed state
  Arms: E4: CG400549 960mg
Drug: Placebo 640mg — multiple oral doses of 640 mg placebo (n=2) BID for 5 days (Days 1-5) and a final dose on Day 6 in the fed state
  Arms: P1 Placebo
Drug: Placebo 320mg — multiple oral doses of 320 mg placebo (n=2) QD for 5 days in the fed state
  Arms: P2: Placebo 320mg
Drug: placebo 960 mg — multiple oral doses of 960 mg placebo (n=2) QD for 5 days in the fed state
  Arms: P3 Placebo 640mg
Drug: Placebo 640mg — multiple oral doses of 640 mg placebo (n=2) QD for 5 days in the fed state
  Arms: P4: Placebo 960mg

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of 3 multiple and escalating dose regimens of CG400549 administered orally in healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, 3 cohorts study consisting of a randomised, double-blind, and placebo-controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-55 years, inclusive
* Body Mass Index :19-30 kg/m2, inclusive
* Sex:male
* Other criteria:healthy; non-smoking or smoking ≤ 10 cigarettes/day

Exclusion Criteria:

* Evidence of clinically relevant pathology
* History of bacterial or viral infection requiring treatment with antibiotics or antivirals within 1 month of study
* Presence or history of esophageal or gastroduodenal ulceration within 1 month before screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From Time the ICF is signed until Follow up Visit (15 days after study drug administration)

SECONDARY OUTCOMES:
Pharmacokinetics-tmax(h), Cmax (ng/mL), Auc (0-24), T1/2(h) | Day1 and Day5
  To determine the pharmacokinetics of CG400549 following oral administration of multiple ascending doses of CG400549 in healthy male subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Seonggu Ro, PhD, Study Chair — CrystalGenomics, Inc.
Locations (1):
- PRA International clinical center, Zuidlaren, Netherlands